CLINICAL TRIAL: NCT04884087
Title: Ecological Momentary Assessment of Substance Use in Homeless Youth
Brief Title: EMA of Substance Use in Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Laura Chavez, Senior Research Scientist, Nationwide Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: STUDY00000809
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design (fixed incentive model vs. prize-based model; random assessment 3x vs. 6x per day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EMA, 3x/day, fixed incentive (Experimental): Ecological Momentary Assessment (EMA; Metricwire). Participants randomized to this group will be sent prompts through the EMA app to complete brief EMA survey at 3 random times per day. Participants randomized to this group will earn a fixed bonus/incentive based on completion of the EMA surveys (50-74%=$3; 75-89%=$5; ≥90%=$10) each week.
  Interventions: Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 3x/day; Behavioral: Incentive Structure - fixed
- EMA, 6x/day, fixed incentive (Experimental): Ecological Momentary Assessment (EMA; Metricwire). Participants randomized to this group will be sent prompts through the EMA app to complete brief EMA survey at 6 random times per day. Participants randomized to this group will earn a fixed bonus/incentive based on completion of the EMA surveys (50-74%=$3; 75-89%=$5; ≥90%=$10) each week.
  Interventions: Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 6x/day; Behavioral: Incentive Structure - fixed
- EMA, 3x/day, prize-based incentive (Experimental): Ecological Momentary Assessment (EMA; Metricwire). Participants randomized to this group will be sent prompts through the EMA app to complete brief EMA survey at 3 random times per day. Participants randomized to this group will be rewarded for high survey completion with increasing numbers of "draws" for prizes depending on their level of response each week (50-74%=1 draw, 75-89%=2 draws, ≥90%=3 draws).
  Interventions: Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 3x/day; Behavioral: Incentive Structure - prize based
- EMA, 6x/day, prized-based incentive (Experimental): Ecological Momentary Assessment (EMA; Metricwire). Participants randomized to this group will be sent prompts through the EMA app to complete brief EMA survey at 6 random times per day. Participants randomized to this group will be rewarded for high survey completion with increasing numbers of "draws" for prizes depending on their level of response each week (50-74%=1 draw, 75-89%=2 draws, ≥90%=3 draws).
  Interventions: Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 6x/day; Behavioral: Incentive Structure - prize based

INTERVENTIONS:
Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 3x/day — Participants receive 3 EMA survey prompts daily for the duration of the study.
  Arms: EMA, 3x/day, fixed incentive; EMA, 3x/day, prize-based incentive
Behavioral: Ecological Momentary Assessment (EMA; Metricwire) Prompts 6x/day — Participants receive 6 EMA survey prompts daily for the duration of the study.
  Arms: EMA, 6x/day, fixed incentive; EMA, 6x/day, prized-based incentive
Behavioral: Incentive Structure - fixed — Those assigned to the "fixed" incentive condition will earn a fixed bonus based on EMA completion (50-74%=$3; 75-89%=$5; ≥90%=$10) each week.
  Arms: EMA, 3x/day, fixed incentive; EMA, 6x/day, fixed incentive
Behavioral: Incentive Structure - prize based — Those assigned to the "prize-based" incentive will be rewarded for high survey completion with increasing numbers of "draws" depending on their level of response to EMA prompts each week (50-74%=1 draw, 75-89%=2 draws, ≥90%=3 draws). For each draw, individuals will use the EMA app to "spin the wheel" to see which prize amount they earn. Out of a total of 500 total draws, 50% will be $1, 43.6% will be $3, 6% will be medium prizes ($5), and 0.4% will be a "jumbo" prize ($90).
  Arms: EMA, 3x/day, prize-based incentive; EMA, 6x/day, prized-based incentive

SUMMARY:
The proposed study will provide critical information on Ecological Momentary Assessment (EMA) design characteristics that promote retention in a vulnerable and under-represented population in research-youth experiencing homelessness. The study will use an EMA app to collect substance use, mood, craving, social surroundings, and trauma measures over a 14-day period in youth age 18-24 (n=40) recruited from Star House, a homeless youth drop-in center. Youth will be randomized in 2x2 factorial design (fixed incentive model vs. prize-based model; random assessment 3x vs. 6x per day).

ELIGIBILITY:
Inclusion Criteria:

* currently homeless, defined as lacking a fixed, regular, and adequate nighttime residence.
* report any of the following past-month frequencies of substance use (NIDA ASSIST screen) used in prior EMA studies: a) heavy episodic or "binge" drinking (≥4 drinks per day for women/≥5 drinks for men) ≥2 days per month ; b) marijuana use ≥2 days per week; or c) any illicit drug use.

Exclusion Criteria:

-

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Length of Time | Baseline to end of trial (day 14)
  Total length of time in days using EMA (range: 1-14 days). Higher values represent greater length of time EMA was used.
Percent Completion | Baseline to end of trial (day 14)
  Percent of EMA surveys completed (0-100%). Higher values represent a larger percentage of EMA surveys completed.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chavez, Principal Investigator — Abigail Wexner Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No